CLINICAL TRIAL: NCT04616638
Title: Effects of a Community-Based Resistance Training Intervention on Independent Functional Performance by Adults With Intellectual Disabilities: A Pilot Randomized Clinical Trial
Brief Title: Effects of Guided Exercise on Functional Performance and Independence in Adults With Intellectual Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Iva Obrusnikova, Associate Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1165646-7
Record Dates: First submitted 2020-10-23; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Intellectual Disability; Exercise; Obesity
Keywords: Functional performance; Intellectual disability; Resistance training; Social cognitive theory
MeSH Terms: conditions — Intellectual Disability; Motor Activity; Obesity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT-POWER Intervention (Experimental): Six familiarization sessions and 20 RT-POWER sessions.
  Interventions: Behavioral: Resistance Training for Empowerment (RT-POWER)
- Control Intervention (Active Comparator): Six control familiarization sessions and 20 traditional RT sessions.
  Interventions: Behavioral: A traditional RT intervention

INTERVENTIONS:
Behavioral: Resistance Training for Empowerment (RT-POWER) — The EG intervention was designed using the Social Cognitive Theory and its four sources of self-efficacy to promote a participant's (a) involvement in exercise planning, (b) muscular strength, and (c) independent functional performance. It consisted of three phases, which were adapted from the Self-Determined Learning Model of Instruction (Wehmeyer et al., 2000). This model draws from theory and research on self-management and self-control (Bandura, 1986; Martin et al., 1988). Participants were taught by their coaches how to (a) set a goal to meet fitness needs (Phase 1), (b) make a plan to meet goals (Phase 2), and (c) adjust actions to complete the plan (Phase 3).
  Arms: RT-POWER Intervention
Behavioral: A traditional RT intervention — The control intervention also consisted of a three-phase instructional process. Consistent with traditional RT interventions (ACSM, 2009), the coaches rather than the participants, were the primary agents for goal-setting, exercise planning, goal attainment monitoring, and readjusting of the exercise plan. Neither the visual activity schedules nor the system of least-to-most prompts was used in this intervention.
  Arms: Control Intervention

SUMMARY:
Adults with intellectual disabilities (ID) have significantly lower levels of fitness compared to the general population. The health benefits of enhanced muscular strength in the general population are well established. In adults with ID, increased muscular strength levels are positively associated with improved aerobic capacity and performance of functional tasks. A concerted effort has been made to design and evaluate resistance training (RT) interventions aimed at increasing muscular strength in adults with ID. While the findings are encouraging, the small number of published studies, missing or poorly described theoretical frameworks or familiarization protocols that guided the RT interventions, and compromised methodological quality raise questions about the actual effects of these interventions and warrant further investigation. The primary purpose of this study is to design and pilot test the effects of an innovative community-based multi-component RT program, Resistance Training for Empowerment (RT-POWER). The primary aim of RT-POWER is to improve muscular strength and independent functional performance in adults with ID. The trial is guided by the SCT theoretical framework. Adults with ID will be randomly allocated to either an experimental group (EG) or a control group (CG). The EG will receive the RT-POWER intervention and the CG will receive an RT intervention traditionally used with the general population. Stage 1 will consist of six familiarization sessions (2 per week for 3 weeks) and Stage 2 will consist of 20 RT sessions (2 per week for 10 weeks). Five hypotheses will be tested: (a) The EG will demonstrate significantly greater increases on the chest-press and leg-press one-repetition maximum (1-RM) tests from baseline to Week 15 compared with the CG; (b) The EG will demonstrate significantly greater increases on the plank test from baseline to Week 15 compared with the CG; (c) The EG will demonstrate significantly greater increases on the six-minute walk test (6MWT) from baseline to Week 15 compared with the CG; (d) The EG will demonstrate significantly greater decreases on the stair climb functional test (SCFT) from baseline to Week 15 compared with the CG; and (e) The EG will demonstrate significantly greater increases in the percentage of steps performed correctly and independently of four RT exercise tasks from baseline to Week 15 compared with the CG.

DETAILED DESCRIPTION:
Participants:

At least 24 participants will be recruited through three disability organizations (two suburban and one urban), all providing transition services, supported employment, and day activity programs for adults with ID. The disability organizations will mail a flyer promoting the study, a screening questionnaire, and consent forms to all parents or legal guardians of adults with ID who the program directors believe met the inclusion criteria.

Exercise Setting:

The study will take place in the fitness-center portion of a large YMCA.

Interventions:

Each intervention will proceed in two stages. Stage 1 - RT-POWER Intervention. The EG will receive six familiarization sessions that promote all four sources of SE. The coaches will first explain terms commonly used in RT using visuals of a model applying the terms during exercise, manipulatives, and live demonstrations in the gym. Two technology-enhanced instructional strategies, a visual activity schedule (VAS) and a video-enhanced system of least-to-most prompting (SLMP), will be utilized to teach participants to correctly and independently perform the four equipment-based RT exercise tasks (chest press, leg press, seated row, and military press) later included in Stage 2. In the investigators' previous work, each exercise task was task analyzed into the specific component steps needed for successful performance. The VAS will be presented to participants via the First Then Visual Schedule HD app (FTVS) on an iPad with a 20cm LED display and wireless headphones. In each familiarization session, participants will retrieve an iPad, headphones, and an exercise log from their coach. After a 10-min warm-up and stretching period, they will complete one set of 10 or 12 repetitions at 50-60% of 1-RM for that exercise task estimated from the baseline measurements. The exercise tasks and the number of repetitions will be counterbalanced across sessions. Both the VAS and the video prompts were pilot tested, and content validity, relevance, and readability of the videos were established with the same machines and population in previous studies conducted by the investigators.

Stage 1 - Control Intervention. This stage will include the same exercise setting, exercise tasks, orientation sessions, exercise log, natural cues, procedural script, and praise as described under Stage 1 - RT-POWER Intervention. The same instruction will be used to alert a participant to begin a task, followed by an opportunity to perform the task. If a participant makes a mistake that cannot be ignored (e.g., set a very heavy weight) or takes more than 15 s to complete a step, the coach performs the step for the participant out of her/his view. Neither the VAS nor the SLMP will be provided to CG participants in this stage.

Stage 2 - RT-POWER Intervention. The intervention consists of three phases, which were adapted from the Self-Determined Learning Model of Instruction. Participants will be taught by their coaches how to (a) set a goal to meet fitness needs (Phase 1), (b) make a plan to meet goals (Phase 2), and (c) adjust actions to complete the plan (Phase 3).

Phase 1 involves Setting a Goal. Participants will be first interview by the coaches to identify their specific strengths and instructional needs and communicate preferences, interests, beliefs, and values pertaining to their health, employment, and home living. Additionally, participants will be shown graphed results of their current level of performance on a 20-cm LED iPad via the Goal-Setting Tracker (GST) that was developed by the investigators using Excel and a graphics tool. The GST converts performance data into two types of graphs. The bar graph is used to present continuous data that do not have a predefined maximum value, such as the level of muscular strength and physical function and the time spent in managerial and transitional tasks. The thermometer graph is used to present a task status toward a predefined maximum value, such as the percentage of exercise steps completed correctly and independently. Using the GST on a 20-cm LED iPad, the coaches teach participants the meaning of their levels of performance and how to set goals that are (a) relevant in addressing their muscular strength and functional performance, (b) specific (i.e., including the FITT parameters), (c) measurable, (d) realistic (i.e., difficult yet attainable), and (e) proximal (i.e., attainable in a short term).

Phase 2 will involve Making a Plan. Participants will be taught to determine, implement, and self-monitor an exercise plan to close the gap from their current performance status to their goal. All exercise plans will include the four equipment-based RT exercises taught during the familiarization stage (i.e., chest press, leg press, seated row, and military press) and two floor core-strengthening exercises (i.e., crunches and prone planks). Similar to Stage 1, each session will start with a 10-min warm-up and stretching period. Next, for machine and dumbbell exercises, participants will complete 1-3 sets of 10-12 repetitions at 50-80% of 1RM for that exercise task. For crunches, participants will complete 1-2 sets of 10-20 repetitions at 3 s per each repetition and with arms either by the sides, on the chest, or behind the head to change resistance. For planks, participants will complete 1-2 sets, holding the position as long as they can while trying to improve their old time. The order of exercise tasks and the number of repetitions will be counterbalanced across sessions. Following ACSM guidelines, the coaches will guide participants to focus their exercise plan on (a) increasing intensity (weight, speed, arm position) and/or volume (repetitions, sets, or time) of the RT exercises; (b) increasing or maintaining the percentage of steps of a task that is completed correctly and independently; and (c) decreasing time spent in managerial tasks (i.e., setting/cleaning up equipment) and transitional tasks (i.e., moving between stations). The intensity will be taught and monitored using the adult OMNI-walk/run rating of perceived exertion (RPE) scale, the adult OMNI-elliptical RPE scale, and the adult OMNI-resistance exercise RPE scale. Additionally, the performance of managerial and transitional tasks at each station will be monitored using a stopwatch.

Phase 3 will involve Tracking Progress. To enhance task/goal self-efficacy, participants and their coaches will jointly monitor progress toward goal attainment and evaluate the success of the exercise plan using GST graphs and verbal instruction delivered by the coach. After goal attainment, following the ACSM's principles of progression, new goals will be set, and the whole process will be reset. If necessary, the Reinforcement Inventory for Adults will be used to select rewards for participation in each session or after goal attainment.

Stage 2 - Control Intervention. The control intervention also will consist of a three-phase instructional process. Consistent with traditional personal training, the coaches rather than the participants will be the primary agents for choices, decisions, and actions. In Phase 1, while current levels of performance will be assessed, the results of the assessment will be not shown visually to the participants. The coaches will set goals that are relevant, specific, measurable, realistic, and proximal. Phase 2 will include the same exercise setting, exercises, session structure, exercise log, natural cues, procedural script, and praise described under the Stage 2 - RT-POWER Intervention. Coaches will design the exercise plan for the participants following the ACSM guidelines; however, the focus of the plan will be on increasing intensity (weight or speed) and/or volume (repetitions or sets) of the RT exercises and not on improving independent functional performance and decreasing the time in managerial and transitional tasks. As in the RT-POWER intervention, the three types of OMNI scale will be used to monitor exercise intensity at each station. Participants will be instructed how to perform exercise tasks with verbal and modeling prompts. Neither the VAS nor the SLMP will be used in this intervention. In Phase 3, the coaches rather than the participant will monitor progress toward goal attainment and evaluate the success of the exercise plan. The coach will set new goals, and the process will be reset. Other than the end-of-the-project reward, no additional rewards will be provided for participation in each session or after goal attainment.

Procedures:

Prior to the baseline assessments and the first intervention session, participants will receive one or two 70-min orientation sessions. Participants will be brought to the YMCA in sizes of four. The four participants will participate in the exercise program and setting during the same time period, but their start times will be staggered. The same coach and research assistant will work with the participant. The same investigators will perform the assessments.

Treatment Fidelity and Social Validity:

The study will emphasize four key areas of treatment fidelity (i.e., establishment, assessment, evaluation, and reporting). Procedural fidelity checks will be performed for all sessions using two fidelity checklists (i.e., one for each group). A trained research assistant who also will be in charge of video recording will note adverse events and missed sessions, and evaluate either in-vivo or indirectly from the recordings a coach's adherence to the prescribed procedures and her/his competence in delivering instruction. Two sets of social validity data will be collected to determine social importance, acceptability, and contextual relevance of the intervention and the procedures. First, the enjoyment of each session will be assessed with the revised Physical Activity Enjoyment Scale (PACES). Second, following the last training session, the coaches, the research assistants, and the participants' job coaches will complete an online social validity questionnaire. The questionnaire consists of 15 seven-point rating items adapted from a well-cited social validity tool measuring intervention acceptability.

Data Analysis:

Descriptive statistics will be computed for each dependent measure and group. The two groups will be examined at baseline for important demographic and clinical characteristics and to verify group homogeneity. Statistical significance of within-group changes between the three measurements will be assessed with paired-samples t-tests. The bivariate Pearson Product Moment correlations will be performed to explore relationships between the baseline performance data and the ID severity, sex, and age of the participants. An intention-to-treat analysis will be conducted with 24 participants to test the study's hypotheses. An analysis of covariance (ANCOVA) will be used to determine the significance (p < .05) of the effects for all outcome measures at 15 weeks between the two groups, with baseline scores used as covariates. Eta squared (η2) will be computed for each effect.

ELIGIBILITY:
Inclusion Criteria:

* an IQ score below 70;
* a chronological age between 18 and 44 years;
* a receptive vocabulary score at or above five years of age;

Exclusion Criteria:

* previous diagnosis of any chronic or co-morbid condition that could affect the performance of the target exercise tasks as assessed by the AHA/ACSM Health/Fitness Facility Preparticipation Screening Questionnaire (ACSM, 2014);
* a record of currently being pregnant or undergoing hormonal replacement or cancer therapy;
* prior or current experience with a similar intervention.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Change in dynamic upper-body and lower-body strength | Change from Baseline to Week 15
  Upper-body and lower-body muscular strength will be measured with the chest-press and the leg-press 1-RM tests (ACSM, 2018), respectively. Each testing session will start with a warm-up set of 6-10 repetitions, with approximately 50% of the estimated resistance. Loads will be estimated with the repetitions-to-fatigue method. Participants will be given 3 attempts. For each attempt, participants will be asked to complete 2 repetitions at the same speed of movement and range of motion. If a participant completes 2 repetitions, the resistance will be increased by 3-10% in the next attempt (or decreased by 3-10% if the first attempt is not successful). This same procedure will be used for the third attempt. The final weight lifted successfully with only one repetition will be recorded to the nearest 5 lb. The rest period will be 3-5 min between the attempts and 5 min between the exercises. Both tests have been used in other clinical trials with adults with ID (Shields et al., 2008).
Change in static trunk strength | Change from Baseline to Week 15
  The prone plank test will measure static trunk strength (ACSM, 2018). After taking shoes off, the participants will be asked to assume the forearm plank position with elbows in contact with the ground, the humerus forming a perpendicular line to the horizontal plane, and the forearms in the neutral position with hands directly in front of the elbows. The timer will start once participants assume a rigid anatomical body position so that only their forearms and toes supported the body. Participants will hold this position as long as possible, and the test will be terminated when the participants voluntarily stop the test, fail to maintain the position, or report ill effect from the test. The total time to hold the position will be measured to the nearest 0.01 s. The best of two trials (30 s between trials to rest) will be used for analysis. The test is a valid and reliable measure for evaluating trunk strength in both younger and older adults (Bohannon et al., 2018).
Change in cardiopulmonary functional capacity | Change from Baseline to Week 15
  Two measures of functional performance were used in this study. The Six-Minute Walk Test (6MWT; American Thoracic Association, 2002) is a submaximal field test of cardiopulmonary functional capacity for activities of daily living (Enright & Sherrill, 1998). The test will be performed using a 50-ft course in the gym. Participants will be instructed to walk as fast as possible for 6 min without running or jogging. During the first lap, a research assistant will walk behind the participant, and then provide standardized encouragement every minute (Casey et al., 2012). The distance walked in 6 min will be measured to the nearest cm. The 6MWT is a reliable (ICC = .96) and a valid test for assessment of cardiorespiratory fitness in adults with mild to severe ID, with strong relationships with VO2 peak and isometric leg strength (Guerra-Balic et al., 2015).
Change in functional mobility | Change from Baseline to Week 15
  The Stairs Climb Functional Test (SCFT; Nightingale et al., 2014) assesses ability to ascend and descend a flight of stairs and lower extremity strength, power, and balance. Participants will be instructed to as quickly as possible ascend, turn, and descend 10 stairs (about 25 cm deep and 16.5 cm high) using any method of traversing the stairs but to take one step at a time and not use the handrails for support. The total time to ascend and descend stairs will be measured to the nearest 0.01 s. The best of three trials (30 s between trials to rest) will be used for analysis. The SCFT is a valid measure of functional mobility in adults with different diagnoses (Nightingale et al., 2014).
Change in performance of RT exercise tasks | Change from Baseline to Week 15
  The performance of four RT exercise tasks (i.e., chest press, leg press, seated row, and military press) will be assessed. A Sony Handycam camcorder will be used to record performance of each exercise task. To observe and code exercise performance, Obrusnikova et al. (2020) and Obrusnikova et al. (2019) developed a coding manual for the four exercise tasks following guidelines proposed by Yoder and Symons (2010). According to the coding manual, a participant's response was considered correct if the performed step conformed to the description in the task analysis (quality), was initiated within 8 s of the exercise directive or completion of the previous step in the task sequence (latency), and was completed within 15 s (duration). The coding manual was piloted and used in previous studies with adults with ID (Obrusnikova et al., 2020; Obrusnikova et al., 2019). To ensure coding reliability, inter-observer agreement (IOA) checks will be completed for all observational data.

CONTACTS AND LOCATIONS:
Overall Officials: Iva Obrusnikova, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- [Background] Cowley PM, Ploutz-Snyder LL, Baynard T, Heffernan K, Jae SY, Hsu S, Lee M, Pitetti KH, Reiman MP, Fernhall B. Physical fitness predicts functional tasks in individuals with Down syndrome. Med Sci Sports Exerc. 2010 Feb;42(2):388-93. doi: 10.1249/MSS.0b013e3181b07e7a. PMID 19927019
- [Background] Bouzas S, Martinez-Lemos RI, Ayan C. Effects of exercise on the physical fitness level of adults with intellectual disability: a systematic review. Disabil Rehabil. 2019 Dec;41(26):3118-3140. doi: 10.1080/09638288.2018.1491646. Epub 2018 Oct 9. PMID 30301367
- [Background] Obrusnikova I, Novak HM, Cavalier AR. The Effect of Systematic Prompting on the Acquisition of Five Muscle-Strengthening Exercises by Adults With Mild Intellectual Disabilities. Adapt Phys Activ Q. 2019 Oct 1;36(4):447-471. doi: 10.1123/apaq.2018-0192. Epub 2019 Sep 13. PMID 31521057
- [Background] Obrusnikova I, Cavalier AR, Novak HM, Blair AE. The Effect of Systematic Prompting on the Acquisition of Two Muscle-Strengthening Exercises by Adults with Moderate Disabilities. J Behav Educ. 2020 Sep;29(3):584-605. doi: 10.1007/s10864-019-09328-7. Epub 2019 May 14. PMID 33737797
- [Background] Wehmeyer ML, Palmer SB, Agran M, Mithaug DE, Martin JE. Promoting causal agency: The self-determined learning model of instruction. Exceptional Children. 2000;66(4):439-53. doi: 10.1177/001440290006600401
- [Background] Latham GP, Locke EA. Enhancing the benefits and overcoming the pitfalls of goal setting. Organizational Dynamics. 2006;35(4):332. doi: 10.1016/j.orgdyn.2006.08.008.
- [Background] Bandura A, Simon KM. The role of proximal intentions in self-regulation of refractory behavior. Cognitive Therapy and Research. 1977;1(3):177. doi: 10.1007/BF01186792
- [Background] Robertson RJ. Perceived exertion for practitioners: rating effort with the OMNI picture system. Champaign, IL: Human Kinetics; 2004.
- [Background] Mays RJ, Goss FL, Schafer MA, Kim KH, Nagle-Stilley EF, Robertson RJ. Validation of adult omni perceived exertion scales for elliptical ergometry. Percept Mot Skills. 2010 Dec;111(3):848-62. doi: 10.2466/05.06.PMS.111.6.848-862. PMID 21319623
- [Background] Strecher VJ, Seijts GH, Kok GJ, Latham GP, Glasgow R, DeVellis B, Meertens RM, Bulger DW. Goal setting as a strategy for health behavior change. Health Educ Q. 1995 May;22(2):190-200. doi: 10.1177/109019819502200207. PMID 7622387
- [Background] Perepletchikova F, Kazdin AE. Treatment integrity and therapeutic change: Issues and research recommendations. Clinical Psychology: Science and Practice. 2005;12(4):365-83. doi: 10.1093/clipsy.bpi045.
- [Background] Motl RW, Dishman RK, Saunders R, Dowda M, Felton G, Pate RR. Measuring enjoyment of physical activity in adolescent girls. Am J Prev Med. 2001 Aug;21(2):110-7. doi: 10.1016/s0749-3797(01)00326-9. PMID 11457630
- [Background] Elliott SN, Treuting MVB. The behavior intervention rating scale: Development and validation of a pretreatment acceptability and effectiveness measure. Journal of School Psychology. 1991;29(1):43-51. doi: 10.1016/0022-4405(91)90014-I.
- [Background] Altman DG, Machin D, Bryant T, Gardner MJ. Statistics with confidence. 2nd ed. London: BMJ Books; 2000
- [Background] American College of Sports Medicine. ACSM's health-related physical fitness assessment manual. 5th ed. Philadelphia, PA: Wolters Kluwer; 2018
- [Background] Shields N, Taylor NF, Dodd KJ. Effects of a community-based progressive resistance training program on muscle performance and physical function in adults with Down syndrome: a randomized controlled trial. Arch Phys Med Rehabil. 2008 Jul;89(7):1215-20. doi: 10.1016/j.apmr.2007.11.056. PMID 18586124
- [Background] Bohannon RW, Steffl M, Glenney SS, Green M, Cashwell L, Prajerova K, Bunn J. The prone bridge test: Performance, validity, and reliability among older and younger adults. J Bodyw Mov Ther. 2018 Apr;22(2):385-389. doi: 10.1016/j.jbmt.2017.07.005. Epub 2017 Jul 25. PMID 29861239
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Enright PL, Sherrill DL. Reference equations for the six-minute walk in healthy adults. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1384-7. doi: 10.1164/ajrccm.158.5.9710086. PMID 9817683
- [Background] Casey AF, Wang X, Osterling K. Test-retest reliability of the 6-minute walk test in individuals with Down syndrome. Arch Phys Med Rehabil. 2012 Nov;93(11):2068-74. doi: 10.1016/j.apmr.2012.04.022. Epub 2012 May 7. PMID 22575394
- [Background] Guerra-Balic M, Oviedo GR, Javierre C, Fortuno J, Barnet-Lopez S, Nino O, Alamo J, Fernhall B. Reliability and validity of the 6-min walk test in adults and seniors with intellectual disabilities. Res Dev Disabil. 2015 Dec;47:144-53. doi: 10.1016/j.ridd.2015.09.011. Epub 2015 Sep 29. PMID 26426514
- [Background] Nightingale EJ, Pourkazemi F, Hiller CE. Systematic review of timed stair tests. J Rehabil Res Dev. 2014;51(3):335-50. doi: 10.1682/JRRD.2013.06.0148. PMID 25019658